CLINICAL TRIAL: NCT06824753
Title: Effect Of Postoperative Pump Blood Administration On Erythrocyte Suspension Requirement And Coagulation Parameters İn Cardiopulmonary Bypass Surgery
Brief Title: Postoperative Use Of Pump Blood İn Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed E Aydin, Assoc Prof, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/186
Record Dates: First submitted 2024-10-11; First posted 2025-02-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cardio-pulmonary Bypass
Keywords: Autologous blood transfusion; ROTEM
MeSH Terms: interventions — Oxygenators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous transfusion group (Active Comparator)
  Interventions: Other: oxygenator and tubing set blood transfusion
- Control Group (No Intervention)

INTERVENTIONS:
Other: oxygenator and tubing set blood transfusion — blood from the oxygenator and tubing set was collected into a 1000 cc Ringer lactate bag, originally used as the pump's priming solution, under sterile conditions using a roller pump
  Arms: autologous transfusion group

SUMMARY:
In our study, the impact of administering autologous blood remaining in the cardiopulmonary bypass system during coronary artery bypass surgeries will be evaluated using the ROTEM device to assess its effect on coagulation parameters. Additionally, the influence of this autologous blood on the need for erythrocyte suspension will be examined, providing insight into its potential role in reducing transfusion requirements in the postoperative period.

Material and Method: The study included 60 patients scheduled for coronary artery bypass graft surgery who met the inclusion criteria. These patients were randomly assigned into two groups: 30 in the study group and 30 in the control group. Following the surgery, all patients were transferred to the intensive care unit under continuous monitoring. In the control group, ROTEM analysis was performed during the first postoperative hour. For the study group, blood from the oxygenator and tubing set was collected into a 1000 cc Ringer lactate bag, originally used as the pump's priming solution, under sterile conditions using a roller pump. The hematocrit levels and the total volume of the collected blood were measured and recorded in milliliters. The study group patients received a 30-minute infusion of this blood at the 1st postoperative hour. ROTEM was performed on the study group after the infusion had concluded.

Postoperative monitoring was carried out at four specific time points: the 4th hour, 24th hour, 48th hour, and upon discharge from the intensive care unit. During this period, the patients' drainage volumes, hemoglobin, hematocrit, leukocyte, and platelet counts were documented. In addition, fluid balance, BUN, and creatinine levels were tracked, along with mechanical ventilator duration and associated parameters. The study concluded with postoperative follow-up, and all collected data were analyzed statistically to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Elective cardiopulmonary bypass surgery
2. Ages 18-70

Exclusion Criteria:

1. Patients not accepting to be included in the study
2. Having kidney disease
3. Having hematological disease
4. Having peripheral artery disease

3- Ejection Fraction < 45% 4- Anticoagulants usage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative need for red blood cell (RBC) transfusion measured by number of RBC units administered | Until the end of the 7th postoperative day
  The primary outcome is the requirement for postoperative red blood cell transfusion. The measurement tool is the number of RBC units transfused, recorded from hospital transfusion records from the end of surgery until the 7th postoperative day.

SECONDARY OUTCOMES:
Incidence of TRALI, TACO, AKI, re-operation, and total drainage amount measured using standard clinical and laboratory criteria | Until the end of the 7th postoperative day
  TRALI: Diagnosed according to the 2019 International Society of Blood Transfusion criteria.
  TACO: Assessed by clinical signs, chest X-ray, and hemodynamic parameters.
  AKI: Evaluated using KDIGO criteria based on serum creatinine and urine output.
  Re-operation: Number of patients requiring surgical re-intervention.
  Drainage amounts: Measured in milliliters from postoperative drains.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennett-Guerrero E, Zhao Y, O'Brien SM, Ferguson TB Jr, Peterson ED, Gammie JS, Song HK. Variation in use of blood transfusion in coronary artery bypass graft surgery. JAMA. 2010 Oct 13;304(14):1568-75. doi: 10.1001/jama.2010.1406. PMID 20940382
- [Result] Paone G, Likosky DS, Brewer R, Theurer PF, Bell GF, Cogan CM, Prager RL; Membership of the Michigan Society of Thoracic and Cardiovascular Surgeons. Transfusion of 1 and 2 units of red blood cells is associated with increased morbidity and mortality. Ann Thorac Surg. 2014 Jan;97(1):87-93; discussion 93-4. doi: 10.1016/j.athoracsur.2013.07.020. Epub 2013 Oct 3. PMID 24094521